CLINICAL TRIAL: NCT00501917
Title: Single Center, Prospective, Randomized, Partly-Double Blinded, Controlled Trial to Assess the Safety and Feasibility of Intracoronary Cell Infusion Mobilized With G-CSF and Darbepoetin and Their Effects on Improvement of Cardiac Function in Patients With Myocardial Infarction: Myocardial Regeneration and Angiogenesis in Myocardial Infarction With G-CSF and Erythropoietin Mobilization and Intra-Coronary Cell Infusion -5-Combination Cytokine Therapy Trial
Brief Title: MAGIC Cell-5-Combicytokine Trial
Acronym: MAGIC Cell-5
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAGIC Cell-5
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-16 (Estimated); Status verified 2007-07

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: G-CSF with/without darbepoetin, peripheral blood stem cell infusion

SUMMARY:
Combination use of darbepoetin and G-CSF will improve left ventricular systolic function in patients with acute myocardial infarction who receive intracoronary infusion of mobilized peripheral blood stem cell in comparison with patient who treated with conventional measures and who received intracoronary infusion of mobilized peripheral blood stem cell by G-CSF alone.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation acute myocardial infarction
* < 80years
* successful revascularization of culprit vessel

Exclusion Criteria:

* uncontrolled congestive heart failure
* uncontrolled myocardial ischemia
* uncontrolled ventricular arrhythmia
* malignancy
* serious hematologic disease
* chronic renal failure

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2007-03; Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
change of left ventricular ejection fraction measured by cardiac MRI | 6, 12, and 24month

SECONDARY OUTCOMES:
wall motion score index exercise capacity BNP | 6,12, 24month

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National Univesity Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang HJ, Yoon EJ, Lee EJ, Kim MK, Suh JW, Park KW, Lee HY, Park KU, Cho YS, Koo BK, Chae IH, Choi DJ, Han KS, Kim HS, Park YB. Cotreatment with darbepoetin and granulocyte colony-stimulating factor is efficient to recruit proangiogenic cell populations in patients with acute myocardial infarction. Cell Transplant. 2012;21(5):1055-61. doi: 10.3727/096368911X627499. Epub 2012 Mar 22. PMID 22449332
- [Derived] Kang HJ, Kim MK, Kim MG, Choi DJ, Yoon JH, Park YB, Kim HS. A multicenter, prospective, randomized, controlled trial evaluating the safety and efficacy of intracoronary cell infusion mobilized with granulocyte colony-stimulating factor and darbepoetin after acute myocardial infarction: study design and rationale of the 'MAGIC cell-5-combination cytokine trial'. Trials. 2011 Feb 7;12:33. doi: 10.1186/1745-6215-12-33. PMID 21299845